CLINICAL TRIAL: NCT00800436
Title: An Open-Label, Two-Part, Multi-Centre, Trastuzumab Dose-Finding Study in Healthy Male Volunteers and HER2 Positive Female Patients
Brief Title: A Dose-Finding Study of Subcutaneous Herceptin (Trastuzumab) in Healthy Male Volunteers and Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP22023
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Results first posted 2016-12-16 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

ARMS (7):
- Part 1: Cohort 1 (Experimental): Healthy male participants will receive Herceptin 6 mg/kg IV on Day 1.
  Interventions: Drug: Herceptin
- Part 1: Cohort 2 (Experimental): Female participants with HER2-positive breast cancer will receive Herceptin 6 mg/kg IV on Day 1.
  Interventions: Drug: Herceptin
- Part 1: Cohort 3 (Experimental): Healthy male participants will receive Herceptin 6 mg/kg SC on Day 1.
  Interventions: Drug: Herceptin
- Part 1: Cohort 4 (Experimental): Healthy male participants will receive Herceptin 10 mg/kg SC on Day 1.
  Interventions: Drug: Herceptin
- Part 1: Cohort 5 (Experimental): Healthy male participants will receive Herceptin SC at an adjusted dose level based on preliminary PK analysis of Cohorts 1, 2, 3, and 4.
  Interventions: Drug: Herceptin
- Part 2: Cohort A (Experimental): Female participants with HER2-positive breast cancer will receive Herceptin SC at the dose level determined in Part 1.
  Interventions: Drug: Herceptin
- Part 2: Cohort B (Experimental): Female participants with HER2-positive breast cancer will receive Herceptin SC at an adjusted dose level based on preliminary PK analysis of Cohort A.
  Interventions: Drug: Herceptin

INTERVENTIONS:
Drug: Herceptin — Herceptin will be administered IV or SC at various dosages (depending upon the cohort to which the participant is assigned) on Day 1.
  Other Names: Trastuzumab

SUMMARY:
This two-part study is designed to select the subcutaneous (SC) dose of Herceptin that results in comparable exposure to intravenous (IV) Herceptin in healthy male participants and in HER2-positive female participants. The study will also assess the safety and tolerability of the SC and IV formulations. In Part 1 of the study, four cohorts will be treated with a single dose of Herceptin as follows: Cohort 1 (6 milligrams per kilogram [mg/kg] IV in healthy male participants); Cohort 2 (6 mg/kg IV in HER2-positive female participants); Cohort 3 (6 mg/kg SC in healthy male participants); Cohort 4 (10 mg/kg SC in healthy male participants). An additional cohort of healthy volunteers (Cohort 5) will be opened if both SC dose levels from Cohorts 3 and 4 result in Herceptin exposures different from the target concentration produced by a single IV dose, or if the variability in pharmacokinetic (PK) parameter values cannot be used to define the target SC dose level. In Part 2 of the study, HER2-positive female participants will receive a single dose of SC Herceptin at the dose level defined in Part 1. Participants from Part 1 are eligible to enter Part 2 provided they receive the second (Part 2) study dose of Herceptin a minimum of 22 days after their first (Part 1) dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Participants (Part 1 only)

  * Males 18 to 45 to years of age
  * Baseline left ventricular ejection fraction (LVEF) greater than (>) 60 percent (%)
* HER2-Positive Females (Parts 1 and 2)

  * Females greater than or equal to (≥) 18 years of age
  * Eastern Cooperative Oncology Group (ECOG) performance status of 0
  * Previous non-metastatic operable primary invasive HER2-positive breast cancer
  * Baseline LVEF >55%

Exclusion Criteria:

* Healthy Participants (Part 1 only)

  * Clinically significant abnormalities in laboratory test results or electrocardiogram
  * History of significant allergies, gastrointestinal, renal, hepatic, cardiovascular, or pulmonary disease
  * History of hypersensitivity or allergic reaction, spontaneous or following drug administration
  * History of cardiac conditions
* HER2-Positive Females (Parts 1 and 2)

  * Metastatic disease
  * Concurrent other malignancy requiring therapy of any modality which may interfere with PK investigations or result in unexpected toxicity
  * Use of Herceptin in previous 5 months
  * Serious cardiac illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- East Bentleigh, Australia
- New Zealand (2):
  - Christchurch
  - Grafton

REFERENCES:
- [Derived] Wynne C, Harvey V, Schwabe C, Waaka D, McIntyre C, Bittner B. Comparison of subcutaneous and intravenous administration of trastuzumab: a phase I/Ib trial in healthy male volunteers and patients with HER2-positive breast cancer. J Clin Pharmacol. 2013 Feb;53(2):192-201. doi: 10.1177/0091270012436560. PMID 23436264

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four participants were counted twice as they were treated in both Cohort 2 and Cohort A.
Groups:
- Part 1: Cohort 1: Healthy male participants received Herceptin 6 milligrams per kilogram (mg/kg) intravenously (IV) on Day 1.
- Part 1: Cohort 2: Female participants with human epidermal growth factor receptor 2 (HER2)-positive breast cancer received Herceptin 6 mg/kg IV on Day 1.
- Part 1: Cohort 3: Healthy male participants received Herceptin 6 mg/kg subcutaneously (SC) on Day 1.
- Part 1: Cohort 4: Healthy male participants received Herceptin 10 mg/kg SC on Day 1.
- Part 1: Cohort 5: Healthy male participants received Herceptin 8 mg/kg SC on Day 1.
- Part 2: Cohort A: Female participants with HER2-positive breast cancer received Herceptin 8 mg/kg SC on Day 1.
- Part 2: Cohort B: Female participants with HER2-positive breast cancer received Herceptin 12 mg/kg SC on Day 1.
Period: Overall Study
Arm/Group | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 1: Cohort 3 | Part 1: Cohort 4 | Part 1: Cohort 5 | Part 2: Cohort A | Part 2: Cohort B
Started | 6 | 6 | 6 | 6 | 6 | 20 | 20
Completed | 6 | 6 | 5 | 5 | 6 | 20 | 20
Not Completed | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who received at least one dose of study medication, whether prematurely withdrawn from the study or not. The "Total" column (n=70) includes 4 female participants who were counted twice as they were treated in both Cohort 2 and Cohort A.
Groups:
- Part 1: Cohort 1: Healthy male participants received Herceptin 6 mg/kg IV on Day 1.
- Part 1: Cohort 2: Female participants with HER2-positive breast cancer received Herceptin 6 mg/kg IV on Day 1.
- Part 1: Cohort 3: Healthy male participants received Herceptin 6 mg/kg SC on Day 1.
- Total: Total of all reporting groups
Arm/Group | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 1: Cohort 3 | Part 1: Cohort 4 | Part 1: Cohort 5 | Part 2: Cohort A | Part 2: Cohort B | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 20 | 20 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.7 (2.58) | 46.2 (5.19) | 25.7 (9.29) | 23.0 (6.16) | 22.0 (4.34) | 50.7 (7.21) | 51.6 (9.04) | 41.2 (14.85)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 6 | 0 | 0 | 0 | 20 | 20 | 46
  Male | 6 | 0 | 6 | 6 | 6 | 0 | 0 | 24

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve Extrapolated to Infinity (AUCinf) of Trastuzumab
Description: AUCinf represents the area under the concentration-time curve of trastuzumab in serum over the time interval from 0 extrapolated to infinity. Values for AUCinf of trastuzumab were derived by non-compartmental analysis across all pharmacokinetic (PK) collections and expressed in days by micrograms per milliliter (days•μg/mL).
Time Frame: Predose (0 hours) and postdose from start of 1.5-hour infusion (1.5 and 3 hours for IV) (6, 8, 12 hours for SC) on Day 1; on Days 2, 3, 5, 8, 15, 22, 43, 85; additionally on Day 10 for SC and Day 35 for IV; and 5 months postdose (up to 5 months overall)
Population: PK Population: All enrolled participants who adhered to the protocol (per protocol basis).
Measure: Mean (Standard Deviation); unit: days•μg/mL
Arm/Group | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 1: Cohort 3 | Part 1: Cohort 4 | Part 1: Cohort 5 | Part 2: Cohort A | Part 2: Cohort B
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 20 | 20
days•μg/mL | 1610 (303) | 1800 (250) | 1350 (320) | 2500 (515) | 1960 (244) | 2090 (638) | 3550 (982)

2. Secondary Outcome: Trough Serum Concentration on Day 22 (CDay22) of Trastuzumab
Description: CDay22 of trastuzumab was derived from the single PK collection on Day 22 and expressed in micrograms per milliliter (μg/mL).
Time Frame: Day 22
Population: PK Population
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 1: Cohort 3 | Part 1: Cohort 4 | Part 1: Cohort 5 | Part 2: Cohort A | Part 2: Cohort B
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 20 | 20
μg/mL | 25.6 (12.1) | 27.5 (7.5) | 31.6 (12.0) | 51.4 (15.8) | 39.4 (5.5) | 37.8 (10.4) | 60.8 (22.0)

3. Secondary Outcome: Maximum Observed Serum Concentration of Trastuzumab (Cmax)
Description: Cmax of trastuzumab was derived across all post-dose PK collections and expressed in μg/mL.
Time Frame: Postdose from start of 1.5-hour infusion (1.5 and 3 hours for IV) (6, 8, 12 hours for SC) on Day 1; on Days 2, 3, 5, 8, 15, 22, 43, 85; additionally on Day 10 for SC and Day 35 for IV; and 5 months postdose (up to 5 months overall)
Population: PK Population
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 1: Cohort 3 | Part 1: Cohort 4 | Part 1: Cohort 5 | Part 2: Cohort A | Part 2: Cohort B
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 20 | 20
μg/mL | 150 (14.4) | 185 (42.9) | 66.8 (11.4) | 102 (17.2) | 82.0 (11.3) | 88.4 (33.3) | 151 (58.6)

4. Secondary Outcome: Time to Maximum Serum Concentration (Tmax) of Trastuzumab
Description: Tmax of trastuzumab was based on the Cmax derived across all post-dose PK collections and expressed in hours.
Time Frame: as for outcome 3
Population: PK Population
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 1: Cohort 3 | Part 1: Cohort 4 | Part 1: Cohort 5 | Part 2: Cohort A | Part 2: Cohort B
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 20 | 20
hours | 1.65 [1.6 to 24.0] | 3.00 [1.55 to 24.0] | 156.00 [95.95 to 216.10] | 132.12 [96.00 to 216.00] | 96.00 [96.00 to 215.98] | 97.13 [47.93 to 216.60] | 96.05 [24.53 to 241.40]

5. Secondary Outcome: Terminal Elimination Half-Life (T1/2) of Trastuzumab
Description: T1/2 of trastuzumab was measured as the time required for trastuzumab concentration to decrease by one-half. T1/2 was derived across all PK collections and expressed in hours.
Time Frame: as for outcome 3
Population: PK Population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 1: Cohort 3 | Part 1: Cohort 4 | Part 1: Cohort 5 | Part 2: Cohort A | Part 2: Cohort B
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 20 | 20
hours | 254 (32.2) | 244 (69.2) | 227 (55.9) | 240 (34.4) | 236 (43.9) | 241 (48.1) | 270 (80.1)

ADVERSE EVENTS:
Time Frame: From Baseline up to 5 months post-dose (up to 5 months overall)
Description: Analysis Population Description: Safety Population
Arm/Group | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 1: Cohort 3 | Part 1: Cohort 4 | Part 1: Cohort 5 | Part 2: Cohort A | Part 2: Cohort B
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 5/6 | 5/6 | 6/6 | 19/20 | 20/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Cohort 1 (N=6) | Part 1: Cohort 2 (N=6) | Part 1: Cohort 3 (N=6) | Part 1: Cohort 4 (N=6) | Part 1: Cohort 5 (N=6) | Part 2: Cohort A (N=20) | Part 2: Cohort B (N=20)
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 1 | 2 | 3
Injection site erythema (General disorders) | 0 | 0 | 1 | 0 | 0 | 4 | 2
Chest pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 2
Injection site discolouration (General disorders) | 0 | 0 | 2 | 0 | 0 | 3 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0
Catheter site haematoma (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2
Infusion related reaction (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Application site inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Application site reaction (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Application site vesicles (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gravitational oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 2 | 2 | 0 | 2 | 12 | 14
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 4 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1
Restless leg syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract Infection (Infections and infestations) | 0 | 0 | 1 | 2 | 1 | 4 | 5
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 3 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 3 | 1
Athralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Joint crepitation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 6 | 2
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysponea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Conjuctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid bleeding (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Scleral hypermia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.